CLINICAL TRIAL: NCT03516968
Title: Treatment of Vitamin D Deficit in Obese Children and Adolescents: an Open Label Randomized Controlled Study Comparing the Efficacy of Two Oral Supplementation Regimens: Monthly Boluses Versus Daily Doses for Correcting Blood Vitamin D Level: OBEVIDOS
Brief Title: Monthly Boluses Versus Daily Doses for Correcting Blood Vitamin D Deficit in Obese Children and Adolescents
Acronym: OBEVIDOS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0148
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Childhood
Keywords: Obesity; Vitamin D deficiency,; supplementation,; Child; Adolescent
MeSH Terms: conditions — Pediatric Obesity; Obesity; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monthly bolus arm (Experimental)
  Interventions: Drug: Monthly bolus of cholecalciferol per os
- Daily arm (Experimental)
  Interventions: Drug: Daily dose of cholecalciferol per os

INTERVENTIONS:
Drug: Monthly bolus of cholecalciferol per os — Bolus therapy: first 50 000 IU and a second 50 IU after 6 weeks
  Arms: Monthly bolus arm
Drug: Daily dose of cholecalciferol per os — Daily substitution, 1200 IU per day (4 drops), for 3 months
  Arms: Daily arm

SUMMARY:
Childhood obesity is one of the most serious public health challenges of the 21st century, with an increasing prevalence over time in developed countries. Overweight and obese children and adolescents are likely to remain so into adulthood and to develop chronic diseases at a young age, such as diabetes and cardiovascular disease.

Obese patients, whether adults or children, are likely to have low serum vitamin D levels due to sequestration and/or volumetric dilution of this fat-soluble vitamin in adipose tissue. Studies have established a link between vitamin D deficiency or insufficiency and chronic diseases such as hypertension, type 2 diabetes and other metabolic problems.

Determining physiological 25(OH)D levels to ensure optimal phosphocalcic metabolism and bone mineralisation requires the use of functional markers: parathyroid hormone (PTH) levels, assessment of the intestinal calcium absorption fraction, assessment of bone mineral density and bone mineral content using absorptiometry.

Vitamin D deficiency leads to malabsorption of calcium and phosphate in the digestive tract, with concentrations, especially of calcium, tending to fall in plasma, resulting in hypersecretion of PTH, which mobilises bone calcium to maintain subnormal blood calcium levels.

Each unit increase in BMI is associated with lower serum vitamin D concentrations: given these low concentrations in this population associated with the risk of developing pathologies, it is important to ensure adequate vitamin D supplementation.

The latest paediatric recommendations recommend, for children aged between 1 and 18 with vitamin D deficiency, a supplement of 2,000 IU/day for at least 6 weeks or a bolus of 50,000 IU once a week for at least 6 weeks.

There are different dosage regimens for the replacement of vitamin D deficiency depending on the country: there is a lack of data on the appropriate dosage and administration regimens for vitamin D supplementation in cases of deficiency, particularly in obese children and adolescents. A prospective, randomised clinical trial will make it possible to define the vitamin D supplementation regimen best suited to increasing serum vitamin D levels in these children and adolescents suffering from obesity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 5 to 18 year-old
* Being obese (BMI >97th percentile, > IOTF 30, for age and gender using the WHO references)
* Patients (parents) having given their informed consent
* Patient having insurance from the national health system

Exclusion Criteria:

Children will be excluded from the study if:

* Symptomatic vitamin D deficiency (tetany, muscular hypotonia, hypocalcaemic seizure)
* Vitamin D supplementation in the 3 months preceding the inclusion visit (V1)
* Signs of rickets at the X-ray (osteopenia and cortical thinning of the long bones, stress fractures, and metaphyseal widening and fraying)
* Chronic disease such as granulomatous conditions, Williams syndrome, or hypothyroidism predisposing to hypocalcaemia or in case of hypercalcaemia (calcium > 2.65 mmol/L), liver/kidney disease, malabsorption diseases;
* Hypercalciuria (urinary Calcium/Creatinine > 0.7 mmol/mmol), calcium nephrolithiasis, hypervitaminosis D (25-(OH)D > 250 nmol/L); nephrocalcinosis;
* Ongoing treatment with anticonvulsants/barbiturates or steroids which increase the catabolism of 25(OH)D;
* Ongoing treatment with thiazides diuretics which reduce urinary excretion of calcium;
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product;
* Pregnancy, breastfeeding;
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant;
* Simultaneous enrolment to another study which could influence the results of the current study;
* Patient under legal protection or deprived of liberty.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reaching the therapeutic target defined as vitamin D (25(OH)D) serum level ≥ 50 nmol/L and < 120 nmol/L | Month 3
  Vitamin D (25OH)D) serum level

SECONDARY OUTCOMES:
calcium dosages | Month 3
  blood safety dosages
phosphore dosages | Month 3
  blood safety dosages
vitamin D (25(OH)D) dosages | Month 3
  blood safety dosages
urinary calcium | Month 3
  urinary safety dosages
creatinin | Month 3
  urinary safety dosages
Treatment compliance | Month 3
  amount of treatment taken (Daily arm: patient diary and weighting of returned treatment at M3. Bolus arm: description of taken ampoules after hospital dosing (number taken, empty or not))
Evaluation of influence of type of skin on study results | Month 3
  assessed a questionnaire
Evaluation of influence of physical activity on study results | Month 3
  assessed by a questionnaire
Evaluation of influence of sun exposure on study results | Month 3
  assessed by a questionnaire
Evaluation of influence of alimentary intakes on study results | Month 3
  assessed by questionnaires
Bone mineral density description (DXA) | Day 1
  Bone mineral density
Evaluation of the PTH variation | Month 3
  PTH serum level
Comparison bone mineral density (DXA) with a preexisting cohort | Day 1
  Bone mineral density (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Carine Villanueva, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - Centre d'Investigation Clinique de LYON - CIC 1407- Groupement Hospitalier Est / Hospices Civils de Lyon, Bron
  - Service d'endocrinologie et métabolisme pédiatrique, Hôpital Femme Mère Enfant, Bron
  - Service d'Endocrinologie Pédiatrique CHU de Clermont-Ferrand, Clermont-Ferrand
  - Centre Médical Infantile de Romagnat, Romagnat

IPD SHARING:
Plan to Share IPD: No